CLINICAL TRIAL: NCT03694028
Title: Neuromuscular and Biomechanical Control of Lower Limb Loading in Individuals With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Vicki Gray, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HP-00072173
Record Dates: First submitted 2018-09-29; First posted 2018-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Stroke; Hemiparesis
Keywords: biomechanical; kinematic; muscle coactivation; torque
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limb Loading (Experimental): This group will be exposed to a sudden unilateral lowering of the supporting surface to induce lateral weight transfer of the paretic limb.
  Interventions: Other: Limb Loading
- Conventional Training (Active Comparator): This group will practice weight shifting and step training that focuses on the paretic limb.
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Limb Loading — Participants will be assigned to one of two interventions. The intervention will occur 3 times a week for six weeks (18 sessions) each session for one hour.
  Arms: Limb Loading
Other: Conventional Training — Participants will be assigned to one of two interventions. The intervention will occur 3 times a week for six weeks (18 sessions) each session for one hour.
  Arms: Conventional Training

SUMMARY:
Stroke is the leading cause of long-term disability in the U.S. Individuals with hemiparesis due to stroke often have difficulty bearing weight on their legs and transferring weight from one leg to the other. The ability to bear weight on the legs is important during functional movements such as rising from a chair, standing and walking. Diminished weight transfer contributes to asymmetries during walking which commonly leads to greater energy expenditure. Moreover, deficits in bearing weight on the paretic leg contribute to lateral instability and are associated with decreased walking speed and increased risk of falling in individuals post-stroke. These functional limitations affect community participation and life quality. Thus, restoring the ability to bear weight on the legs, i.e., limb loading, is a critical goal for rehabilitation post-stroke. The purpose of this research is to identify the impairments in neuromechanical mechanisms of limb loading and determine whether limb loading responses can be retrained by induced forced limb loading.

DETAILED DESCRIPTION:
Stroke is the leading cause of long-term disability in the U.S. Individuals with hemiparesis due to stroke often have difficulty bearing weight on the paretic lower extremity and transferring weight from one leg to the other. Impaired weight transfer and limb loading contribute to lateral instability and are associated with decreased walking speed and increased risk of falling. Consequently, restoring limb loading ability is an important goal for rehabilitation post-stroke. Despite considerable rehabilitation efforts aimed at enhancing paretic limb loading, their effectiveness on improving neuromotor and functional outcomes remains limited possibly due to poorly understood limb loading mechanisms and the reluctance to use the paretic limb. The coordination of neuromuscular actions to regulate loading force during weight acceptance is an important component of functional limb loading. Because altered neuromuscular control is common in persons with stroke, it is possible that these abnormalities may impair limb loading ability. The long-term objective of this project is to develop a mechanism-based framework for designing and testing the effectiveness of novel rehabilitation interventions to enhance lower limb weight transfer and limb loading to improve balance and mobility. This project aims to (1) identify the neuromuscular and biomechanical abnormalities in limb loading responses in individuals post-stroke, (2) determine the underlying mechanisms responsible for the deficits in limb loading, and (3) test the short-term effectiveness of a 6-week perturbation-induced limb load training program on improving limb loading responses and mobility function. The investigators propose to apply a sudden unilateral lowering of the supporting surface to induce lateral weight transfer that forces limb loading. Kinetic, kinematic, and lower extremity muscle activation patterns will be recorded. The investigators expect that, compared to healthy controls, individuals with stroke will show increased muscle co-activation of the knee musculature with decreased knee flexion and torque production, and irregular impact force regulation during loading that will disrupt weight transfer and loading of the paretic limb. Furthermore, the investigators hypothesize that compared to a conventional clinical weight-shift rehabilitation training program, the imposed limb loading group will show greater improvements during voluntary stepping and walking following training. Specifically, the investigators expect the knee muscle co-activation duration will be reduced, with increased knee joint torque, and the paretic single stance/double support time will increase, reflecting improved paretic limb loading ability during gait following training.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis as a result of a stroke greater than 6 months previous to the study if participants with stroke.
* Able to walk 10 meters with or without a walking aid.
* Able to stand unsupported for 5 minutes.

Exclusion Criteria:

* Medical condition precluding participation in regular exercises, such as acute cardiac or respiratory conditions limiting activity and other health conditions significantly impacting the ability to walk beyond the effects of the stroke, such as other neurological conditions or peripheral neuropathies.
* Not able to follow commands.
* Pregnancy by self-report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Gait single stance time asymmetry and duration ratio | Post training at 6 weeks
  single stance time asymmetry and duration ratio
Gait paretic double support/single stance | Post training at 6 weeks
  paretic double support/single stance
Stepping weight transfer time | Post training at 6 weeks
  weight transfer time
Stepping knee angular displacement | Post training at 6 weeks
  knee angular displacement
Stepping peak torque | Post training at 6 weeks
  peak torque

CONTACTS AND LOCATIONS:
Overall Officials: Vicki L Gray, MPT, PhD, Principal Investigator — Assistant Professor
Locations (1):
- PTRS Research Lab, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No